CLINICAL TRIAL: NCT00348647
Title: Can Lower Extremity Overuse Injuries Be Prevented by an Exercise Program Aiming at Muscular Strength, Flexibility and Coordination - a RCT
Brief Title: Prevention of Injuries by an Exercise Program - a RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amager Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2003-1-62
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2006-07-04 (Estimated); Status verified 2004-12

CONDITIONS: Patellofemoral Pain Syndrome; Exertional Lower Leg Pain
Keywords: Prevention; Exercise; Overuse; Anterior knee pain syndrome; Exertional lower leg pain; Prospective; Risk factors; Hip
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Motor Activity

INTERVENTIONS:
Behavioral: physical training program to prevent injuries

SUMMARY:
Overuse injuries are a major concern for physical active individuals. Study hypothesis is that an exercise programme based on known intrinsic risk factors can prevent overuse injuries in soldiers undergoing basic military training.

DETAILED DESCRIPTION:
PURPOSE: Overuse injuries are a major concern for physical active individuals engaged in endurance type activities. This is especially true for soldiers during basic military training or subjects with a sedentary lifestyle taking up exercise to prevent disease, as they are vulnerable for sustaining an overuse injury. Contradictory to traumatic injuries, little is known about the prevention of overuse injuries using a training program. This study evaluates the preventive effect of a training program based on known intrinsic risk factors for the occurrence of anterior knee pain and shin pain in soldiers undergoing basic military training. We also evaluate the effect on physical performance.

METHODS: From December 2004 - March 2006 1000 soldiers undergoing basic military training divided into 24 platoons are cluster randomised into a prevention-training (PRE) group or a placebo-training (PLA) group. The PRE group will perform exercises based on known intrinsic risk factors namely strength, flexibility and coordination of the lower extremity, while the PLA group will perform exercises for the upper body. Both programmes consists of 5 exercises and will be performed 3 times a week during a 12 weeks period. All subjects will prospectively be examined by the same observer, who will be blinded to the allocation.

OUTCOME: primary outcome: reduction in anterior knee pain and shin pain.

ELIGIBILITY:
Inclusion Criteria:

* Basic military training in the Royal Danish Guards.
* Passed military medical board.

Exclusion Criteria:

* Injury before start of intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900
Dates: Start 2004-12; Study Completion 2006-03

PRIMARY OUTCOMES:
reduction in anterior knee pain
reduction in shin pain

SECONDARY OUTCOMES:
reduktion in overuse injuries
physical performance

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Brushoj, MD, Principal Investigator — Amager Hospital DK-2300 Amager